CLINICAL TRIAL: NCT02178319
Title: Randomized Clinical Trial Comparing Laparoscopic and Open Esophagogastric Devascularization and Splenectomy for Portal Hypertension
Brief Title: Laparoscopic Versus Open Devascularization for Portal Hypertension, a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: portal hypertension
Record Dates: First submitted 2014-06-19; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Portal Hypertension; Liver Cirrhosis
Keywords: portal hypertension; Randomized clinical trial; laparoscopic; open
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis | interventions — Conversion to Open Surgery; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- open group (Active Comparator): the patients under go the open esophagogastric devascularization and splenectomy
  Interventions: Procedure: open surgical procedure
- laparoscopic group (Experimental): the patients under go the laparoscopic esophagogastric devascularization and splenectomy
  Interventions: Procedure: laparoscopic surgical procedure

INTERVENTIONS:
Procedure: open surgical procedure — open esophagogastric devascularization and splenectomy will perform as surgical procedure in the patients
  Arms: open group
Procedure: laparoscopic surgical procedure — laparoscopic esophagogastric devascularization and splenectomy will perform as surgical procedure in the patients
  Arms: laparoscopic group

SUMMARY:
Many patients with portal hypertension require surgical treatment each year,and Hassab's operation, or esophagogastric devascularization and splenectomy, is an elective procedure. In recent years,laparoscopic esophagogastric devascularization and splenectomy has been used to treat portal hypertension. However, the potential benefits remain to be demonstrated in the context of a randomized trial. In this study, 120 patients will randomize equally receiving laparoscopic or open esophagogastric devascularization and splenectomy. Inclusion criteria included: platelet count < 50×109/ml, esophageal and gastric varices revealed, agreeing the informed consent. PerioperativeOutcomes are: technical success, blood loose and infusion during the operation, recurrent varicose veins on gastroscopy examination, patterns of reflux on duplex ultrasound examination, complications, platelet and liver function variation, length of hospital stay. Follow-up will last 5 years, and gastroscopy and ultrasonic will perform at 3 months, 1 year, 3 years, and 5 years. Further more, this study was proved by the ethical committee of second hospital of Xi'an jiaotong university.

ELIGIBILITY:
Inclusion Criteria:

* The cause of portal hypertension was cirrhosis
* Platelet count < 50×109/ml
* Esophageal and gastric varices revealed
* Agreeing the informed consent.

Exclusion Criteria:

* Thrombosis present in portal vein preoperatively
* Accompany with liver cancer
* Operation procedure is laparoscopy converse to open
* Patients disagree with the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-06; Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
recurrence | 5 years
  gastroesophageal varices recurrence rate

SECONDARY OUTCOMES:
operation time | 1 day
  Duration of surgical procedure

OTHER OUTCOMES:
blood loss during surgical procedure | 1 day
blood transfusion during surgical procedure | 1 day
Number of Participants with Serious and Non-Serious Adverse Events | 4 weeks
  record all kind of postoperative complications in each patient
rebleeding | 1 day
  record rebleeding time in each bleeding patient
cost of hospitalization | 4 weeks
survival | 5 years
  record the time of death and the death reason
length of hospital stay | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery , Second Afﬁliated Hospita l, Xi'an Jiaotong Universi ty School of Medicine, Xi'an, China